CLINICAL TRIAL: NCT00849446
Title: Validity and Reliability of an Activity Monitor in Persons With a Cerebrovascular Accident
Status: Completed | Type: Observational
Sponsor: University College of Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Other Study IDs: ARTESIS-DepG-2009-1
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-02

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke | interventions — Fitness Trackers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Activity monitoring in CVA patients
  Interventions: Device: Activity monitor (SenseWear Pro armband)
- Activity monitoring in healthy persons
  Interventions: Device: Activity monitor (SenseWear Pro armband)

INTERVENTIONS:
Device: Activity monitor (SenseWear Pro armband) — Activity monitoring during specific physical activities such as walking at different speeds
  Other Names: Sensewear

SUMMARY:
Background:Accelerometry has only recently been introduced in clinical stroke research. However, whether accelerometry is a valid and reliable tool in stroke needs to be established. From literature becomes clear that existing accelerometers show shortages at patients with stroke because of the specific deficits that these patients have.

Purpose: The aim of this study is to investigate the validity and test-retest reliability of the SenseWear Pro armband as an objective measurement of physical activity in chronic stroke patients.

Patients and Methods Subjects: Fifteen patients and fifteen healthy subjects will be included in the study following written informed consent. The following demographic and clinical data were recorded: age, gender, height, length, medication use, self-reported handedness, Edinburgh Handedness Inventory, Rivermead Gross Function, Functional Ambulation Categories, medical and surgical history.

Methods: During one test session the subjects had to carry out an amount of activities according to a standardised protocol existing of lying down, sitting, standing, walking, step exercise and cycling. These activities are presenting activities of daily living.

Measures:Subjects wear on both arms a SenseWear Pro Armband. De data from these measuring devices will be compared with the data retrieved from 2 Yamax pedometers and the ergospirometry device. The outcome measures are: counts, heartbeat, oxygen used, energy expenditure, METabolic equivalent, time lying down.

DETAILED DESCRIPTION:
Evaluation of the SenseWear Pro Armband to assess physical activity in individuals with chronic stroke

Background:

Accelerometry has only recently been introduced in clinical stroke research. However, whether accelerometry is a valid and reliable tool in stroke needs to be established. From literature becomes clear that existing accelerometers show shortages at patients with stroke because of the specific deficits that these patients have.

Purpose:

The aim of this study is to investigate the validity and test-retest reliability of the SenseWear Pro armband as an objective measurement of physical activity in chronic stroke patients.

Patients and Methods Subjects Fifteen patients and fifteen healthy subjects will be included in the study following written informed consent. The following demographic and clinical data were recorded: age, gender, height, length, medication use, self-reported handedness, Edinburgh Handedness Inventory, Rivermead Gross Function, Functional Ambulation Categories, medical and surgical history.

Methods During one test session the subjects had to carry out an amount of activities according to a standardised protocol existing of lying down, sitting, standing, walking, step exercise and cycling. These activities are presenting activities of daily living.

Measures:

Subjects wear on both arms a SenseWear Pro Armband. De data from these measuring devices will be compared with the data retrieved from 2 Yamax pedometers and the ergospirometry device. The outcome measures are: counts, heartbeat, oxygen used, energy expenditure, METabolic equivalent, time lying down.

ELIGIBILITY:
Inclusion criteria:

* an ischemic or hemorrhagic stroke
* stroke onset less than 3 months
* score 3 or more Functional Ambulation Categories
* age < 80 years
* ability to cycle independently
* written authorisation on the informed consent

Exclusion criteria:

* serious other diseases which might have an influence on carrying out the standardised activities
* cannot understand and carry out simple instructions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Fifteen patients and fifteen healthy subjects will be included in the study following written informed consent. The following demographic and clinical data were recorded: age, gender, height, length, medication use, self-reported handedness, Edinburgh Handedness Inventory, Rivermead Gross Function, Functional Ambulation Categories, medical and surgical history.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Total energy expenditure (kcal)during selected physical activities | measurement at 1 time point

SECONDARY OUTCOMES:
Number of steps | measurement at 1 time point

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Antwerp, Edegem, Antwerp, Belgium